CLINICAL TRIAL: NCT01619085
Title: An Open-label Extension Trial of the Long Term Safety of Oral BIBF 1120 in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: Extension Trial of the Long Term Safety of BIBF 1120 in Patients With Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1199.33; 2011-002766-21 (EudraCT Number)
Record Dates: First submitted 2012-06-06; First posted 2012-06-14 (Estimated); Results first posted 2018-07-26 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-02

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — nintedanib

ARMS (1):
- All subjects (Experimental): patient to receive a capsule containing Nintedanib twice a day
  Interventions: Drug: Nintedanib

INTERVENTIONS:
Drug: Nintedanib — Nintedanib twice a day
  Other Names: BIBF 1120

SUMMARY:
The aim of this extension trial is to assess the long-term safety of BIBF 1120 treatment in patients with Idiopathic Pulmonary Fibrosis who have completed one year treatment and the follow up period in the double-blind phase III placebo controlled parent trials (1199.32 and 1199.34), who wish to continue treatment with BIBF 1120.

ELIGIBILITY:
Inclusion criteria:

1. Signed Informed Consent consistent with International Conference on Harmonisation-Good Clinical Practices (ICH-GCP) and local laws prior to trial participation.
2. Patients from trials 1199.32 or 1199.34 who completed the 52 weeks treatment period and performed the follow-up visit.

Exclusion criteria:

1. Aspartate aminotransferase (AST), Alanine aminotransferase (ALT) > 1.5 fold Upper Limit of Normal (ULN) (Patients who completed the parent trial with transaminase values > 1.5 fold ULN but < 3 fold ULN are considered eligible)
2. Bilirubin > 1.5 fold ULN
3. Bleeding risk
4. Planned major surgery within the next 3 months, including lung transplantation, major abdominal or major intestinal surgery.
5. New major thrombo-embolic events developed after completion of the parent trial.
6. Time period > 12 weeks between Visit 9 of the parent trial and Visit 2 of this study.
7. Usage of any investigational drug after completion of the parent trial or planned usage of a specific investigational drug during the course of this trial.
8. A disease or condition which in the opinion of investigator may put the patient at risk because of participation in this trial or limit the patients' ability to participate in this trial.
9. Alcohol or drug abuse which in the opinion of the investigator would interfere with trial participation.
10. Pregnant women or women who are breast feeding or of child bearing potential not using two effective methods of birth control (one barrier and one highly effective non-barrier) for at least 1 month prior to Visit 2 and/or not committing to using it until 3 months after end of treatment.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 752 (Actual)
Dates: Start 2012-06-06 (Actual); Primary Completion 2017-07-05 (Actual); Study Completion 2021-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (172):
- United States (37):
  - Jasper Summit Research, LLC, Jasper, Alabama
  - Pulmonary Associates, Phoenix, Arizona
  - University of California, Los Angeles, California
  - University of California, San Francisco, California
  - Sansum Clinic, Santa Barbara, California
  - Stanford University Medical Center, Stanford, California
  - University of California, Torrance, California
  - Western Connecticut Medical Group, Danbury, Connecticut
  - Pulmonary Assoc of Stamford, Stamford, Connecticut
  - Cleveland Clinic, Weston, Florida
  - Georgia Clinical Research, Austell, Georgia
  - University of Chicago, Chicago, Illinois
  - Via Christi Clinic, PA, Wichita, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - Minnesota Lung Center, Minneapolis, Minnesota
  - The Lung Research Center, LLC, Chesterfield, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Pulmonary and Critical Care Associates, Albany, New York
  - Jamaica Hospital Medical Center, Jamaica, New York
  - New York Presbyterian Hospital, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - ID Clinical Research, LTD, Toledo, Ohio
  - The Oregon Clinic, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - FDC Seifer PLC Pulmonary, Shelbyville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Metroplex Pul and Sleep Ctr, McKinney, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - Vermont Lung Center, Colchester, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Lynchburg Pulmonary Associates, Lynchburg, Virginia
  - University of Wisconsin, Madison, Wisconsin
- Australia (4):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Repatriation General Hospital, Concord, New South Wales
  - Frankston Hospital, Frankston, Victoria
  - Alfred Hospital, Melbourne, Victoria
- Belgium (4):
  - ULB Hopital Erasme, Brussels
  - Brussels - UNIV UZ Brussel, Brussels
  - UZ Leuven, Leuven
  - Yvoir - UNIV UCL de Mont-Godinne, Yvoir
- Canada (2):
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
- Instituto Nacional del Tórax, Santiago, Chile
- China (11):
  - Peking University People's Hospital, Beijing
  - Beijing Friendship Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Xiangya Hospital, Central South University, Changsha
  - West China Hospital, Chengdu
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Zhongshan Hospital Fudan University, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - General Hospital of Shenyang Military Region, Shenyang
  - Xijing Hospital, Xi'an
  - General Hospital of Ningxia Medical University, Yinchuan
- Czechia (3):
  - Thomayer Hospital, Prague
  - University Hospital Na Bulovce, Prague, Prague
  - Masaryk Hospital, Usti nad Labem, Ústí nad Labem
- Finland (2):
  - HYKS Keuhkosairauksien tutkimusyksikkö, Helsinki
  - Mehiläinen Kielotie, Vantaa, Vantaa
- France (13):
  - HOP Avicenne, Bobigny
  - HOP Bocage, Dijon
  - HOP Calmette, Lille
  - HOP Louis Pradel, Lyon
  - HOP Nord, Marseille
  - HOP Arnaud de Villeneuve, Montpellier
  - HOP Pasteur, Nice
  - HOP Européen G. Pompidou, Paris
  - HOP Bichat, Paris
  - HOP Tenon, Paris
  - HOP Maison Blanche, Reims
  - HOP Pontchaillou, Rennes
  - HOP Larrey, Toulouse
- Germany (15):
  - CIMS Studienzentrum Bamberg GmbH, Bamberg
  - Helios Klinikum Emil von Behring, Berlin
  - Evangelische Lungenklinik Berlin, Buch
  - Universitätsklinikum Carl Gustav Carus Dresden, Coswig
  - Klinik Donaustauf, Donaustauf
  - Ruhrlandklinik, Westdeutsches Lungenzentrum am Universitätsklinikum Essen gGmbH, Essen
  - Universitätsklinikum Freiburg, Freiburg/Breisgau
  - Universitätsklinikum Gießen und Marburg GmbH, Giessen
  - Universitätsmedizin Greifswald, Greifswald
  - Pneumologisches Forschungsinstitut an der LungenClinic Grosshansdorf GmbH, Großhansdorf
  - Universitätsklinikum Heidelberg, Heidelberg
  - Lungenfachklinik Immenhausen, Immenhausen
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Klinikum der Universität München - Campus Großhadern, München
  - Universitätsklinikum Münster, Münster
- Greece (3):
  - Athens Hospital of Chest Diseases "Sotiria", Athens
  - University Hospital of Heraklion, University Pulmonology Cl, Heraklion
  - General University Hospital of Larissa, Larissa
- India (6):
  - Mehta Hospital & Cardiopulmonary Care Centre, Ahmedabad
  - Chest & Maternity Center, Bangalore
  - Asthma Bhawan, Jaipur
  - National Allergy Asthma Bronchitis Institute, Kolkata, Kolkata
  - P.D. Hinduja National Hospital, Mumbai
  - Jahingir Clinical Development Centre, Pune
- Mater Misericordiae University Hospital, Dublin, Ireland
- Israel (2):
  - Rabin Medical Center Beilinson, Petah Tikva
  - Kaplan Medical Center, Rehovot
- Italy (10):
  - Osp. Clin. SS. Anunziata, Chieti Scalo
  - Ospedale "G.B. Morgagni - L. Pierantoni" ausl forli, Forlì
  - Osp. S. Giuseppe Fatebenefratelli, Milan
  - Università di Modena e Reggio Emilia, Modena
  - A.O. San Gerardo di Monza, Monza
  - Università Federico II, Napoli
  - Università degli Studi Padova, Padua
  - Ospedale di Cisanello, Pisa
  - Pol. Universitario Tor Vergata, Roma
  - A.O.U. Senese Policlinico Santa Maria alle Scotte, Siena
- Japan (25):
  - Nagoya University Hospital, Aichi, Nagoya
  - Tosei General Hospital, Aichi, Seto
  - Ogaki Municipal Hospital, Gifu, Ogaki
  - National Hospital Organization Himeji Medical Center, Himeji, Hyogo
  - Kobe City Medical Center General Hospital, Hyogo, Kobe
  - Ibarakihigashi National Hospial, Ibaraki, Naka-gun
  - Toranomon Hospital Kajigaya, Kanagawa, Kawasaki
  - Kanagawa Cardiovascular and Respiratory Center, Kanagawa, Yokohama
  - Tohoku University Hospital, Miyagi, Sendai
  - Tenri Hospital, Nara, Tenri
  - Kindai University Hospital, Osaka, Osaka-sayama
  - Saitama Cardiovascular and Respiratory Center, Saitama, Kumagaya
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Sakai, Osaka
  - Jichi Medical University Hospital, Tochigi, Shimotsuke
  - Tokushima University Hospital, Tokushima, Tokushima
  - Tokyo Medical and Dental University, Tokyo, Bunkyo-ku
  - Nippon Medical School Hospital, Tokyo, Bunkyo-ku
  - Fukujuji Hospital, Tokyo, Kiyose
  - Toranomon Hospital, Tokyo, Minato-ku
  - The Jikei University Hospital, Tokyo, Minato-ku
  - Toho University Omori Medical Center, Tokyo, Ota-ku
  - JR Tokyo General Hospital, Tokyo, Shibuya-ku
  - Tokyo Medical University Hospital, Tokyo, Shinjuku-ku
  - Center Hospital of the National Center for Global Health and Medicine, Tokyo, Shinjuku-ku
  - Tottori University Hospital, Tottori, Yonago
- Instituto Nacional de Enfermedades Respiratorias Ismael Cosío Villegas, Mexico City, Mexico
- Netherlands (3):
  - OLVG, locatie Oosterpark, Amsterdam
  - St. Antonius ziekenhuis, locatie Nieuwegein, Nieuwegein
  - Erasmus Medisch Centrum, Rotterdam
- Portugal (5):
  - CHUC - Centro Hospitalar e Universitário de Coimbra, EPE, Coimbra
  - CHLC, EPE - Hospital de Santa Marta, Lisbon
  - Centro Hospitalar Lisboa Norte Hospital Pulido Valente, Lisbon
  - Centro Hospitalar Universitário São João,EPE, Porto
  - Centro Hospitalar de Vila Nova de Gaia, Vila Nova de Gaia
- Scientific Research Institute of Pulmonology, Saint Petersburg, Russia
- South Korea (6):
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Soonchunhyang University Hospital Seoul, Seoul
  - The Catholic University of Korea, Yeouido St.Mary's Hospital, Seoul
- Spain (4):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Nuestra Señora de Valme, Seville
- Turkey (Türkiye) (5):
  - Ankara Universitesi Tip Fakultesi, Ankara
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi, Istanbul
  - Yedikule Gog. Hst. EAH, Istanbul
  - Ege Universitesi T.F., Izmir
  - Dr.Suat Seren EAH, Izmir
- United Kingdom (8):
  - Aberdeen Royal Infirmary, Aberdeen
  - Queen Elizabeth Hospital, Birmingham
  - Birmingham Heartlands Hospital, Birmingham
  - St James's University Hospital, Leeds
  - Aintree University Hospital, Liverpool
  - Royal Brompton Hospital, London
  - Churchill Hospital, Oxford
  - Southmead Hospital, Westbury on Trym

REFERENCES:
- [Derived] Crestani B, Huggins JT, Kaye M, Costabel U, Glaspole I, Ogura T, Song JW, Stansen W, Quaresma M, Stowasser S, Kreuter M. Long-term safety and tolerability of nintedanib in patients with idiopathic pulmonary fibrosis: results from the open-label extension study, INPULSIS-ON. Lancet Respir Med. 2019 Jan;7(1):60-68. doi: 10.1016/S2213-2600(18)30339-4. Epub 2018 Sep 14. PMID 30224318
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a prospective, open-label extension trial in which patients with Idiopathic pulmonary fibrosis (IPF), who had completed 52 weeks of treatment and the follow-up period in the randomised, double-blind, placebo-controlled parent trials 1199.32(NCT01335464)/.34(NCT01335477) and who needed access to nintedanib outside of the discontinued parent trials 1199.35(NCT01170065)/.187(NCT01979952).
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Total (1199.32/.34/.35/.187): For patients participated in parent trials 1199.32/.34 (both were randomized, placebo-controlled): patients were to receive continuous dosing of soft gelatin capsules of nintedanib (orally) 150 milligrams (mg) twice daily (bid) in this study unless they had reduced the dose to 100 mg bid trial drug (nintedanib or placebo) in the parent trial; patients receiving 100 mg bid trial drug at the end of the parent trial could receive either nintedanib 100 mg bid or nintedanib 150 mg bid in this study. The daily nintedanib dose for such patients was decided at baseline visit based on discussion between the patient and the investigator. After unblinding of the parent trials, patients randomized to placebo in parent trials, who reduced the dose to 100 mg bid in the parent trial, could increase the dose to nintedanib 150 mg bid in this study. The dose could also be increased to 150 mg at a later time point if medically justified in this study. For patients participated in parent trials 1199.35/.187 (1199.35: open label; 1199.187: randomized placebo-control): patients were to receive the same daily dosage of soft gelatin capsules of nintedanib (orally) as in the parent trials (100 mg bid or 150 mg bid) in this study. In this study, patients were treated with nintedanib until they met one of the discontinuation criteria. Potential reasons for treatment discontinuation include impaired liver function, recurrence of diarrhoea, and progression of idiopathic pulmonary fibrosis.
Period: Overall Study
Arm/Group | Total (1199.32/.34/.35/.187)
Started | 752
Treated | 751
Completed ('completed' stands for not prematurely discontinued from trial medication) | 227
Not Completed | 525
Not completed — Adverse Event | 231
Not completed — Protocol Violation | 4
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 45
Not completed — Other than specified | 96
Not completed — Not treated | 1
Not completed — Death | 145

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The data set consisted of all patients who were dispensed trial medication and were documented to have taken at least one dose, and had participated in 1199.32/.34 parent trials.
Groups:
- Total (1199.32/.34): This group included patients originated from parent trials 1199.32/.34.
  For patients participated in parent trials 1199.32/.34, they were to receive continuous dosing of soft gelatin capsules of nintedanib (orally) 150 milligrams (mg) twice daily (bid) in this study unless they had reduced the dose to 100 mg bid trial drug (nintedanib or placebo) in the parent trial; patients receiving 100 mg bid trial drug at the end of the parent trial could receive either nintedanib 100 mg bid or nintedanib 150 mg bid in this study. The daily nintedanib dose for such patients was decided at baseline visit based on discussion between the patient and the investigator. After unblinding of the parent trials, patients randomized to placebo in parent trials, who reduced the dose to 100 mg bid in the parent trial, could increase the dose to nintedanib 150 mg bid in this study. The dose could also be increased to 150 mg at a later time point if medically justified in this study.
  In this study, patients were treated with nintedanib until they met one of the discontinuation criteria. Potential reasons for treatment discontinuation include impaired liver function, recurrence of diarrhoea, and progression of idiopathic pulmonary fibrosis.
Arm/Group | Total (1199.32/.34)
Number analyzed (Participants) | 734
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.2 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147
  Male | 587
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 214
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 431
  More than one race | 0
  Unknown or Not Reported | 86

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events (AEs)
Description: This is the measure for percentage of patients with adverse events (AEs) observed during the trial. The incidence of adverse events (% of patients) over the course of the trial, including the incidence of serious AEs, AEs leading to discontinuation, and fatal AEs are presented.
Time Frame: From first drug administration until end of treatment period + 28 days, in total up to 56.3 months plus 28 days.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of patients (%)
Arm/Group | Total (1199.32/.34)
Number analyzed (Participants) | 734
Percentage of patients (%)
  Any AEs | 98.5
  AEs leading to discontinuation of trial drug | 42.6
  Serious AEs | 68.9
  Fatal AEs | 23.8

ADVERSE EVENTS:
Time Frame: From first drug administration in this study until 28 days after the last drug, up to 7.5 years.
Description: Treated set (TS) [and TS35; TS187]: The data set consisted of all patients who were dispensed trial medication and were documented to have taken at least one dose, and had participated in 1199.32/.34 [in 1199.35 for TS35; in 1199.187 for TS187] parent trials. TS (from 1199.32/.34), TS35 (from .35), and TS187 (from .187) are all used to reported the AEs.
Groups:
- Placebo (1199.32/.34): Patients in this group are those who were randomized to placebo arm in parent trials 1199.32/.34 and were treated with 100 milligrams or 150 milligrams of nintedanib orally twice daily in this study.
- Nintedanib 150 Bid (1199.32/.34): Patients in this group are those who were randomized to 150 milligrams nintedanib twice daily (bid) arm in the parent trials 1199.32/.34 and were treated with 100 milligrams or 150 milligrams of nintedanib orally twice daily in this study.
- Placebo (1199.187): Patients in this group are those who were randomized to placebo arm in parent trial 1199.187 and were treated with 150 milligrams or 100 milligrams of nintedanib twice daily in this study.
- Nintedanib 100 Bid (1199.35): Patients in this group are those who were participated in the parent trial 1199.35 and were treated with 100 milligrams of nintedanib twice daily (bid) in this study.
- Nintedanib 150 Bid (1199.35/.187): Patients in this group are those who were treated with 150 milligrams (mg) of nintedanib twice daily (bid) in this study and were participated in parent trial 1199.35 plus those who were randomized to 150 mg nintedanib bid arm in the parent trial 1199.187 and were treated with 150 mg or 100 mg nintedanib bid in this study.
- Total (1199.35/.187): This group included patients originated from parent trials 1199.35/.187. For patients participated in parent trials 1199.35/.187, they were to receive the same daily dosage of soft gelatin capsules of nintedanib (orally) as in the parent trials (100 milligrams (mg) twice daily (bid) or 150 mg bid) in this study.
  In this study, patients were treated with nintedanib until they met one of the discontinuation criteria. Potential reasons for treatment discontinuation include impaired liver function, recurrence of diarrhoea, and progression of idiopathic pulmonary fibrosis.
Arm/Group | Total (1199.32/.34) | Placebo (1199.32/.34) | Nintedanib 150 Bid (1199.32/.34) | Placebo (1199.187) | Nintedanib 100 Bid (1199.35) | Nintedanib 150 Bid (1199.35/.187) | Total (1199.35/.187) | Total (1199.32/.34/.35/.187)
All-Cause Mortality (participants affected / at risk) | 182/734 | 78/304 | 104/430 | 0/7 | 0/2 | 0/8 | 0/17 | 182/751
Serious Adverse Events (participants affected / at risk) | 509/734 | 208/304 | 301/430 | 0/7 | 0/2 | 1/8 | 1/17 | 510/751
Other Adverse Events (participants affected / at risk) | 671/734 | 281/304 | 390/430 | 3/7 | 1/2 | 2/8 | 6/17 | 677/751
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total (1199.32/.34) (N=734) | Placebo (1199.32/.34) (N=304) | Nintedanib 150 Bid (1199.32/.34) (N=430) | Placebo (1199.187) (N=7) | Nintedanib 100 Bid (1199.35) (N=2) | Nintedanib 150 Bid (1199.35/.187) (N=8) | Total (1199.35/.187) (N=17) | Total (1199.32/.34/.35/.187) (N=751)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Acute coronary syndrome (Cardiac disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 6 | 1 | 5 | 0 | 0 | 0 | 0 | 6
Angina pectoris (Cardiac disorders) | 5 | 3 | 2 | 0 | 0 | 0 | 0 | 5
Angina unstable (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 9 | 6 | 3 | 0 | 0 | 0 | 0 | 9
Atrial flutter (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 3
Cardiac arrest (Cardiac disorders) | 4 | 3 | 1 | 0 | 0 | 0 | 0 | 4
Cardiac failure (Cardiac disorders) | 12 | 6 | 6 | 0 | 0 | 0 | 0 | 12
Cardiac failure acute (Cardiac disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 7 | 1 | 6 | 0 | 0 | 0 | 0 | 7
Cardio-respiratory arrest (Cardiac disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Conduction disorder (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cor pulmonale (Cardiac disorders) | 8 | 1 | 7 | 0 | 0 | 0 | 0 | 8
Cor pulmonale chronic (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 9 | 2 | 7 | 0 | 0 | 0 | 0 | 9
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 6 | 2 | 4 | 0 | 0 | 0 | 0 | 6
Mitral valve incompetence (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 4 | 1 | 3 | 0 | 0 | 0 | 0 | 4
Myocardial ischaemia (Cardiac disorders) | 5 | 3 | 2 | 0 | 0 | 0 | 0 | 5
Myocarditis (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Right ventricular failure (Cardiac disorders) | 5 | 3 | 2 | 0 | 0 | 0 | 0 | 5
Tachycardia (Cardiac disorders) | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 3
Porokeratosis (Congenital, familial and genetic disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Deafness (Ear and labyrinth disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Vestibular disorder (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Thyroid mass (Endocrine disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Amaurosis fugax (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Blindness transient (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 3
Dry age-related macular degeneration (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Glaucoma (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Optic ischaemic neuropathy (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Panophthalmitis (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Periorbital fat herniation (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Posterior capsule opacification (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Retinal artery occlusion (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Retinal detachment (Eye disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Retinal vein occlusion (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Anal fistula (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 10 | 5 | 5 | 0 | 0 | 0 | 0 | 10
Duodenal ulcer (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 1 | 3 | 0 | 0 | 0 | 0 | 4
Haematochezia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 4 | 1 | 3 | 0 | 0 | 0 | 0 | 4
Ileus (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Inguinal hernia (Gastrointestinal disorders) | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 4
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Obstruction gastric (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 4 | 1 | 3 | 0 | 0 | 0 | 0 | 4
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pancreatitis necrotising (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Protein-losing gastroenteropathy (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Asthenia (General disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Chest discomfort (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 11 | 3 | 8 | 0 | 0 | 0 | 0 | 11
Complication associated with device (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Condition aggravated (General disorders) | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 3
Death (General disorders) | 3 | 0 | 3 | 0 | 0 | 0 | 0 | 3
Disease progression (General disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Gait disturbance (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Malaise (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 4 | 2 | 2 | 0 | 0 | 0 | 0 | 4
Oedema peripheral (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 4 | 1 | 3 | 0 | 0 | 0 | 0 | 4
Sudden death (General disorders) | 5 | 1 | 4 | 0 | 0 | 0 | 0 | 5
Bile duct stone (Hepatobiliary disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Biliary colic (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 3
Cholecystitis acute (Hepatobiliary disorders) | 6 | 4 | 2 | 0 | 0 | 0 | 0 | 6
Cholelithiasis (Hepatobiliary disorders) | 9 | 4 | 5 | 0 | 0 | 1 | 1 | 10
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Hepatitis (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Liver disorder (Hepatobiliary disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Liver injury (Hepatobiliary disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Biliary sepsis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 12 | 2 | 10 | 0 | 0 | 0 | 0 | 12
Bronchitis bacterial (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Cholecystitis infective (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Enteritis infectious (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Hepatitis A (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Herpes simplex encephalitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Infected cyst (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 7 | 4 | 3 | 0 | 0 | 0 | 0 | 7
Intervertebral discitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 9 | 4 | 5 | 0 | 0 | 0 | 0 | 9
Oral fungal infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Paraspinal abscess (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Peritonitis (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Pleural infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Pneumonia (Infections and infestations) | 99 | 40 | 59 | 0 | 0 | 0 | 0 | 99
Pneumonia bacterial (Infections and infestations) | 5 | 1 | 4 | 0 | 0 | 0 | 0 | 5
Pneumonia influenzal (Infections and infestations) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Postoperative abscess (Infections and infestations) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Pulmonary mycosis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Respiratory syncytial virus infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 13 | 8 | 5 | 0 | 0 | 0 | 0 | 13
Respiratory tract infection bacterial (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Rhinovirus infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 8 | 3 | 5 | 0 | 0 | 0 | 0 | 8
Septic shock (Infections and infestations) | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 3
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Spinal cord abscess (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Tinea capitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Tuberculosis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 7 | 1 | 6 | 0 | 0 | 0 | 0 | 7
Urinary tract infection (Infections and infestations) | 4 | 2 | 2 | 0 | 0 | 0 | 0 | 4
Urosepsis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 6 | 4 | 2 | 0 | 0 | 0 | 0 | 6
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 4
Head injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Hypobarism (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Postoperative delirium (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 4 | 3 | 1 | 0 | 0 | 0 | 0 | 4
Road traffic accident (Injury, poisoning and procedural complications) | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 3
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Blood urea increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Body temperature increased (Investigations) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 2
C-reactive protein increased (Investigations) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Fibrin D dimer increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Glycosylated haemoglobin increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 5 | 2 | 3 | 0 | 0 | 0 | 0 | 5
Transaminases increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 1 | 3 | 0 | 0 | 0 | 0 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0 | 3 | 0 | 0 | 0 | 0 | 3
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 3
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 3
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 2 | 6 | 0 | 0 | 0 | 0 | 8
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 3 | 0 | 0 | 0 | 0 | 3
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 4 | 3 | 0 | 0 | 0 | 0 | 7
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 4 | 9 | 0 | 0 | 0 | 0 | 13
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 3
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Metastases to eye (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 3
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 3
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pleural neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1 | 4 | 0 | 0 | 0 | 0 | 5
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 2 | 4 | 0 | 0 | 0 | 0 | 6
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 4 | 4 | 0 | 0 | 0 | 0 | 8
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1 | 3 | 0 | 0 | 0 | 0 | 4
Tumour of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Brain hypoxia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Cerebral artery occlusion (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cerebral artery stenosis (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cerebral atrophy (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 3 | 0 | 3 | 0 | 0 | 0 | 0 | 3
Coma (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Encephalopathy (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Lacunar infarction (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Radiculopathy (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Syncope (Nervous system disorders) | 9 | 3 | 6 | 0 | 0 | 0 | 0 | 9
Transient ischaemic attack (Nervous system disorders) | 5 | 2 | 3 | 0 | 0 | 0 | 0 | 5
Completed suicide (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Disorientation (Psychiatric disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Hallucination (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 7 | 3 | 4 | 0 | 0 | 0 | 0 | 7
Anuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Azotaemia (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Glomerulonephritis (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Glomerulonephritis chronic (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Lower urinary tract symptoms (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Obstructive nephropathy (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Prerenal failure (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 5 | 3 | 2 | 0 | 0 | 0 | 0 | 5
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 5 | 3 | 2 | 0 | 0 | 0 | 0 | 5
Genital prolapse (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 15 | 4 | 11 | 0 | 0 | 0 | 0 | 15
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 4 | 0 | 0 | 0 | 0 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 38 | 16 | 22 | 0 | 0 | 0 | 0 | 38
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3 | 0 | 0 | 0 | 0 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 2 | 0 | 0 | 0 | 0 | 4
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 13 | 9 | 4 | 0 | 0 | 0 | 0 | 13
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 153 | 64 | 89 | 0 | 0 | 0 | 0 | 153
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 10 | 3 | 7 | 0 | 0 | 0 | 0 | 10
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 3
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 15 | 6 | 9 | 0 | 0 | 0 | 0 | 15
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 11 | 5 | 6 | 0 | 0 | 0 | 0 | 11
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 17 | 11 | 6 | 0 | 0 | 0 | 0 | 17
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 12 | 3 | 9 | 0 | 0 | 0 | 0 | 12
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 48 | 22 | 26 | 0 | 0 | 0 | 0 | 48
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 2 | 0 | 0 | 0 | 0 | 4
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 35 | 9 | 26 | 0 | 0 | 0 | 0 | 35
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Transurethral prostatectomy (Surgical and medical procedures) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Aortic dissection (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Aortic stenosis (Vascular disorders) | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 3
Arterial thrombosis (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 0 | 3 | 0 | 0 | 0 | 0 | 3
Hypotension (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Peripheral artery occlusion (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Shock (Vascular disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Thrombosis (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Blood loss anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Prosthetic cardiac valve thrombosis (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Vascular stent stenosis (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Congestive hepatopathy (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hepatic mass (Hepatobiliary disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Complicated appendicitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Large intestine infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Post procedural fever (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Imaging procedure abnormal (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cutaneous T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cyanosis (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Total (1199.32/.34) (N=734) | Placebo (1199.32/.34) (N=304) | Nintedanib 150 Bid (1199.32/.34) (N=430) | Placebo (1199.187) (N=7) | Nintedanib 100 Bid (1199.35) (N=2) | Nintedanib 150 Bid (1199.35/.187) (N=8) | Total (1199.35/.187) (N=17) | Total (1199.32/.34/.35/.187) (N=751)
Abdominal pain (Gastrointestinal disorders) | 63 | 32 | 31 | 0 | 0 | 0 | 0 | 63
Abdominal pain upper (Gastrointestinal disorders) | 48 | 21 | 27 | 0 | 0 | 0 | 0 | 48
Constipation (Gastrointestinal disorders) | 57 | 26 | 31 | 0 | 0 | 0 | 0 | 57
Diarrhoea (Gastrointestinal disorders) | 514 | 213 | 301 | 2 | 0 | 0 | 2 | 516
Nausea (Gastrointestinal disorders) | 146 | 70 | 76 | 0 | 0 | 0 | 0 | 146
Vomiting (Gastrointestinal disorders) | 89 | 36 | 53 | 0 | 0 | 0 | 0 | 89
Asthenia (General disorders) | 39 | 18 | 21 | 0 | 0 | 0 | 0 | 39
Chest pain (General disorders) | 39 | 15 | 24 | 0 | 0 | 0 | 0 | 39
Fatigue (General disorders) | 68 | 32 | 36 | 0 | 0 | 0 | 0 | 68
Oedema peripheral (General disorders) | 50 | 17 | 33 | 0 | 0 | 0 | 0 | 50
Pyrexia (General disorders) | 42 | 15 | 27 | 0 | 0 | 0 | 0 | 42
Bronchitis (Infections and infestations) | 145 | 54 | 91 | 0 | 0 | 0 | 0 | 145
Lower respiratory tract infection (Infections and infestations) | 40 | 14 | 26 | 0 | 0 | 0 | 0 | 40
Respiratory tract infection (Infections and infestations) | 47 | 15 | 32 | 0 | 0 | 0 | 0 | 47
Rhinitis (Infections and infestations) | 39 | 18 | 21 | 0 | 0 | 0 | 0 | 39
Upper respiratory tract infection (Infections and infestations) | 109 | 38 | 71 | 0 | 0 | 0 | 0 | 109
Weight decreased (Investigations) | 123 | 63 | 60 | 0 | 0 | 0 | 0 | 123
Decreased appetite (Metabolism and nutrition disorders) | 104 | 58 | 46 | 0 | 0 | 0 | 0 | 104
Arthralgia (Musculoskeletal and connective tissue disorders) | 49 | 18 | 31 | 0 | 0 | 0 | 0 | 49
Back pain (Musculoskeletal and connective tissue disorders) | 57 | 28 | 29 | 0 | 0 | 0 | 0 | 57
Dizziness (Nervous system disorders) | 48 | 23 | 25 | 0 | 0 | 0 | 0 | 48
Headache (Nervous system disorders) | 42 | 18 | 24 | 0 | 0 | 0 | 0 | 42
Cough (Respiratory, thoracic and mediastinal disorders) | 166 | 66 | 100 | 0 | 0 | 0 | 0 | 166
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 118 | 48 | 70 | 0 | 0 | 1 | 1 | 119
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 80 | 32 | 48 | 0 | 0 | 0 | 0 | 80
Hypertension (Vascular disorders) | 49 | 23 | 26 | 1 | 0 | 0 | 1 | 50
Cataract (Eye disorders) | 26 | 8 | 18 | 0 | 0 | 1 | 1 | 27
Influenza (Infections and infestations) | 35 | 11 | 24 | 0 | 1 | 0 | 1 | 36
Nasopharyngitis (Infections and infestations) | 152 | 62 | 90 | 0 | 0 | 0 | 0 | 152
Pneumonia (Infections and infestations) | 45 | 19 | 26 | 0 | 0 | 0 | 0 | 45
Myalgia (Musculoskeletal and connective tissue disorders) | 21 | 10 | 11 | 0 | 0 | 1 | 1 | 22
Anxiety (Psychiatric disorders) | 26 | 17 | 9 | 0 | 0 | 0 | 0 | 26
Insomnia (Psychiatric disorders) | 36 | 14 | 22 | 0 | 0 | 0 | 0 | 36
Productive cough (Respiratory, thoracic and mediastinal disorders) | 36 | 12 | 24 | 0 | 0 | 0 | 0 | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-03-28): https://cdn.clinicaltrials.gov/large-docs/85/NCT01619085/Prot_002.pdf
  • Statistical Analysis Plan (2017-07-25): https://cdn.clinicaltrials.gov/large-docs/85/NCT01619085/SAP_003.pdf